CLINICAL TRIAL: NCT03903809
Title: A Phase 3, Randomized, Open-Label, Active-Controlled, Multicenter, Non-Inferiority Study to Evaluate the Efficacy and Safety of Pegol-Sihematide for Anemia in Patients With Non-Dialysis-Dependent Chronic Kidney Disease
Brief Title: Study of the Efficacy and Safety of Pegol-Sihematide for Anemia in Patients With NDD-CKD
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS-20039-301
Record Dates: First submitted 2019-03-04; First posted 2019-04-04 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Non-Dialysis-Dependent Chronic Kidney Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HS-20039 Pegol-Sihematide (Experimental): Pegol-Sihematide's starting dose of 0.025 milligram per kilogram (mg/kg) administered subcutaneously (SC) once every 4 weeks (Q4W) for a total of 13 doses
  Interventions: Drug: Pegol-Sihematide
- ReHuman Erythropoietin Injection (Active Comparator): ESPO(Recombinant Human Erythropoietin Injection) ESPO's starting dose was 6000 IU per week
  Interventions: Drug: ESPO

INTERVENTIONS:
Drug: Pegol-Sihematide — Participants received Pegol-Sihematide by subcutaneous injection once every 4 weeks. The starting dose was 0.04 milligram per kilogram (mg/kg) and was adjusted throughout the study to maintain a hemoglobin target range of 10.0-12.0 grams per deciliter (g/dL).
  Other Names: HS-20039
  Arms: HS-20039 Pegol-Sihematide
Drug: ESPO — Participants received ESPO by subcutaneous injection weekly. The starting dose was 6000 IU and was adjusted according to the instruction to maintain a hemoglobin target range of 10.0-12.0 grams per deciliter (g/dL).
  Other Names: Recombinant Human Erythropoietin Injection
  Arms: ReHuman Erythropoietin Injection

SUMMARY:
The primary objective of this study is to evaluate the safety and efficacy of Pegol-Sihematide, as compared with recombinant human erythropoietin injection (CHO Cell), ESPO, in anemia treatment in patients with non-dialysis-dependent chronic kidney disease.

DETAILED DESCRIPTION:
This is a phase 3, randomized, multicenter, open-label, active-controlled, non-inferiority trial to evaluate the safety and efficacy of Pegol-Sihematide versus ESPO. Study included a period of 4 weeks for screening, 16 weeks for dose adjustment, 8 weeks for evaluation, and 28 weeks for extensional treatment period. Eligible patients were centrally allocated in a 2:1 ratio to receive Pegol-Sihematide subcutaneously once every 4 weeks, starting at 0.04 mg per kilogram of body weight, or ESPO once every 1 week or 2 weeks, starting dose of 6000 IU per week. Doses of both drugs were adjusted to achieve and maintain hemoglobin levels between 10.0 and 12.0 g per deciliter for 52 weeks or more. The primary efficacy end point was the mean change from the baseline hemoglobin level to the mean level during the evaluation period; non-inferiority was established if the lower limit of the two-sided 95% confidence interval was -1.0 g per deciliter or higher. Cardiovascular safety was evaluated on the basis of an adjudicated composite end point.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following inclusion criteria to be eligible for participation in this study:

  1. Males or females ≥ 18 years of age.
  2. Females of child-bearing potential who are sexually active had to be willing to practice a highly effective method of birth control for at least 4 weeks prior to randomization, and had to be willing to continue contraception until at least 4 weeks after the last dose of study treatment.
  3. CKD with an estimated glomerular filtration rate < 60 mL/min/1.73m2 using Collaborative Group on Epidemiology of Chronic Kidney Diseases (CKD-EPI) formula within 4 weeks prior to randomization, and was not expected to begin dialysis for at least 12 weeks.
  4. The patient was not received any erythropoiesis stimulating agents (ESAs) treatment within 12 weeks prior to randomization. And two consecutive hemoglobin values ≥ 6.0 g/dL and < 10.0 g/dL within 4 weeks prior to randomization.
  5. At least one transferrin saturation (TSAT) ≥ 20% or one serum ferritin (SF) level ≥ 100 ng/ml within 4 weeks prior to randomization. At least one serum folate level and vitamin B12 level ≥ lower limit of normal during the 4 weeks prior to randomization.
  6. Patient was informed of the investigational nature of the study and had given written, informed consent in accordance with institutional, local, and national guidelines.

Exclusion Criteria:

* Subjects who meet any of the following exclusion criteria are not to be enrolled in this study:

  1. Females who were pregnant or breast-feeding.
  2. Red blood cell (RBC) or whole blood transfusion within 12 weeks prior to randomization.
  3. Known intolerance to any ESA, parenteral iron supplementation, or PEGylated molecule.
  4. Known hematological disease (including but not limited to myelodysplastic syndrome, hematological malignancy, hemoglobinopathy, pure red cell aplasia, hemolytic syndromes, coagulation disorder, etc.) or cause of anemia other than renal disease（e.g. gastrointestinal bleeding or hookworm disease for stool occult blood positive，etc.）.
  5. Known autoimmune diseases（e.g. rheumatoid arthritis, systemic lupus erythematosus, anti-neutrophil cytoplasmic antibody related vasculitis, etc.）.
  6. Obvious infection occurred within 4 weeks prior to randomization，per investigator's clinical judgment.
  7. Chronic, uncontrolled, or symptomatic inflammatory disease，per investigator's clinical judgment.
  8. Uncontrolled or symptomatic secondary hyperparathyroidism，per investigator's clinical judgment.
  9. Poorly controlled hypertension within 4 weeks prior to randomization, per investigator's clinical judgment.
  10. Chronic congestive heart failure (New York Heart Association Class III~IV).
  11. Active hepatitis or any of the following check exceptions: ALT≥ 2 × upper limit of normal (ULN), AST≥ 2 × upper limit of normal (ULN), DBIL≥ 2 × upper limit of normal (ULN).
  12. A positive test for HIV antibody.
  13. Significant symptoms or diseases within 6 months prior to randomization，and the investigator judged that these diseases or symptoms may affect evaluation or follow-up.
  14. Currently receiving and requiring long-term immunosuppressive therapy.
  15. Tumor malignancy（non-melanoma skin cancer and carcinoma in situ that have been resected are excluded）.
  16. Expected survival less than 12 months.
  17. Elective surgery during the study.
  18. Expected conception within 4 weeks after the end of the study treatment.
  19. The subject has participated in other clinical trial within the 12 weeks prior to randomization and throughout the trial period.
  20. Have any other condition or prior therapy that, in the investigator's opinion, would make the subject unsuitable for the study, or unable or unwilling to comply with the study procedures.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The mean change from the baseline hemoglobin level to the mean level during the evaluation period | Week 17-24
  The primary efficacy end point is the mean change from the baseline hemoglobin level to the mean level during the evaluation period. The baseline hemoglobin value is the value on the day of randomization. The mean hemoglobin during the evaluation period was calculated as the mean of all available hemoglobin values during that period. Hemoglobin measurements will be performed at baseline and thereafter every 2 weeks (for the dose adjustment and the evaluation periods). Efficacy will be also assessed as the mean change from baseline in hemoglobin levels during 4-week intervals.

SECONDARY OUTCOMES:
The mean change from the baseline hemoglobin level to the mean level at each visit | Week 0-52
  The mean change from the baseline hemoglobin level to the mean level at each visit point. Hemoglobin measurements will be performed at every 2 weeks during the dose adjustment period (0-16 weeks) and the evaluation period (17-24 weeks) , and every 4 weeks during the extended period (25-52 weeks).
The proportion of patients with hemoglobin within the target range of 10.0 to 12.0 g/dL during the evaluation period | Week 17-24
  The proportion of patients achieving a response (hemoglobin maintain in 10.0 to 12.0 g/dL during the previous 4 weeks), will be measured during the evaluation period.
The mean dose of patients with Pegol-Sihematide achieving a target hemoglobin range during the evaluation period | Week 17-24
  The mean dose of patients with Pegol-Sihematide will be calculated for achieving a target hemoglobin range (10.0 to 12.0 g/dL) during the evaluation period.
First time for patients achieving a response to hemoglobin during any treatment periods | Week 0-52
  First time for patients achieving a response (hemoglobin increase in ≥ 1.0 g/dL) during any trial periods, including the dose adjustment period (0-16 weeks), the evaluation period (17-24 weeks) and the extended period (25-52 weeks).
First time for patients achieving a target hemoglobin range during any trial periods | Week 0-52
  First time for patients achieving a target hemoglobin range (hemoglobin maintain in 10.0 to 12.0 g/dL or increase in ≥ 1.0 g/dL) during any trial periods, including the dose adjustment period (0-16 weeks), the evaluation period (17-24 weeks) and the extended period (25-52 weeks).

OTHER OUTCOMES:
The SAE of Pegol-Sihematide | Week 0-52
  The incidence of patients who reported serious adverse events (SAE).
The incidence of patients with risk cardiovascular events of Pegol-Sihematide | Week 0-52
  The incidence of patients with risk cardiovascular events, including death, stroke, myocardial infarction and severe congestive heart failure, unstable angina, arrhythmia requiring hospitalization.
The antibody of Pegol-Sihematide | Week 0-52
  The antibody to Pegol-Sihematide is the anti-drug antibodies of the Pegol-Sihematide.

CONTACTS AND LOCATIONS:
Overall Officials: JunqiJunqi Chen, MD, Study Director — The First Affiliated Hospital, Zhejiang University
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Xie J, Yang A, Qiu H, Peng X, Lu W, Huang X, Chen Q, Zhong A, Tang S, Wang Q, Li C, He L, Jia X, Ma A, Wang F, Yu X. Randomized Trial of Pegmolesatide for the Treatment of Anemia in Patients With Nondialysis CKD. Kidney Int Rep. 2024 Dec 6;10(3):720-729. doi: 10.1016/j.ekir.2024.12.002. eCollection 2025 Mar. PMID 40225393